CLINICAL TRIAL: NCT07329439
Title: Comparative Effects of High Intensity and Eccentric Resistance on Squat Strength,Dynamic Balance and Explosive Power Among School Going Basketball Players
Brief Title: Comparative Effects of High Intensity and Eccentric Resistance Among School Going Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0492
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Basketball
Keywords: High intensity resistance training; Eccentric resistance training; Basketball players

STUDY DESIGN:
Intervention Model Description: Randomized control design
Who Masked: Outcomes Assessor
Masking Description: outcome accessors are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 20 participants in group A will receive high intensity resistance training, 8-week duration for significant results. Exercises will be performed at starting 50% of one-repetition maximum (1RM) for hypertrophy and strength gains.
  Interventions: Other: High intensity resistance training
- Group B (Active Comparator): 20 participants in group B will receive eccentric resistance training, 8-week duration for significant results, exercise training three times a week.
  Interventions: Other: Eccentric resistance training

INTERVENTIONS:
Other: High intensity resistance training — group A receive high intensity resistance training, 8-week duration for significant results. Exercises will be performed at starting 50% of one-repetition maximum (1RM) for hypertrophy and strength gains
  Arms: Group A
Other: Eccentric resistance training — Group B receive eccentric resistance training, 8-week duration for significant results, exercise training three times a week.
  Arms: Group B

SUMMARY:
This will be experimental randomized clinical trial conducted in Pakistan sports board, Sacred Heart cathedral high school . Female school going basketball players will be screened for eligibility according to inclusion and exclusion criteria. Informed consent will be obtained from eligible participants. All participants will go through randomization by Online Randomization tool. Information regarding number of groups, number of participants in each group and total number of participants will be entered. This will be a single blinded study in which outcome assessor will be blinded to ensure accuracy and reduce biasness. Sample size according to G power will be 40.

DETAILED DESCRIPTION:
This study purpose is to compare effects of high-intensity and eccentric resistance training on squat strength, dynamic balance, and explosive power among school going basketball players.

This will be experimental randomized clinical trial conducted in Pakistan sports board, Sacred Heart cathedral high school . Female school going basketball players will be screened for eligibility according to inclusion and exclusion criteria. Informed consent will be obtained from eligible participants. All participants will go through randomization by Online Randomization tool. Information regarding number of groups, number of participants in each group and total number of participants will be entered. This will be a single blinded study in which outcome assessor will be blinded to ensure accuracy and reduce biasness. Sample size according to G power will be 40. Group A will receive high intensity resistance training, 8-week duration for significant results. Exercises will be performed at starting 50% of one-repetition maximum (1RM) for hypertrophy and strength gains. Group B will receive eccentric resistance training, 8-week duration for significant results, exercise training three times a week. Training will start at 50% of maximum eccentric force, with adjustments made bi-weekly to maintain this intensity as strength improves. Trainings will be conducted 2-3 times per week includes 3-6 sets of 6-12 repetitions with rest intervals of 30 seconds to 2 minutes. Both groups will be assessed by 1RM squat strength, YBT test and vertical jump test before after training. Objective of this research will be to determine comparative effects of high intensity and eccentric resistance training on squat strength, dynamic balance and power. The data will be analyzed using SPSS version 26 for Windows software. Statistical significance will be set at P = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-18 years
* Female basketball players
* Normal body mass index value
* Must have 6 months basketball experience
* Willingness to complete all study procedures
* Achieve minimum baseline scores in objective physical tests relevant to the study

Exclusion Criteria:

* General health issues
* Ankle sprains
* History of ACL injuries
* Cardiovascular and respiratory disease
* Current involvement in any other research study
* History of major bone injuries in last six months
* Involve in any previous resistance training program

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
1RM squat strength | 8 weeks
  The one-repetition maximum (1RM) test is a widely used strength assessment that measures the maximum amount of weight an individual can lift for a single repetition of a given exercise.This test is typically conducted after a proper warm-up and involves gradually increasing the weight until the participant reaches their maximum lift capacity. The 1RM is a valuable indicator of muscular strength and is commonly utilized in strength training programs.
vertical jump | 8-weeks
  The vertical jump is frequently used as a measurement of lower-body explosive power in the strength and conditioning field. Coaches and researchers consider vertical jump height as one of the essential athletic skills that translate into increased performance in the athlete's respective sport. Vertical jump training is frequently implemented in sports that require explosive movements
Y balance test | 8-weeks
  To perform the Y-Balance Test, an individual stands on one leg and reaches with the other foot to push a sliding box in three directions: anterior (forward), posterolateral (back and to the outside), and posteromedial (back and to the inside), measuring the farthest reach in each direction while maintaining balance. After practice trials, three recorded attempts are made for each direction on each leg.

CONTACTS AND LOCATIONS:
Overall Officials: Masooma Irfan, DPT, Principal Investigator — Riphah International University
Locations (1):
- Sacred Heart Cathedral High School, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva AF, Aghidemand MH, Kharatzadeh M, Ahmadi VK, Oliveira R, Clemente FM, Badicu G, Murawska-Cialowicz E. Effects of High-Intensity Resistance Training on Physical Fitness, Hormonal and Antioxidant Factors: A Randomized Controlled Study Conducted on Young Adult Male Soccer Players. Biology (Basel). 2022 Jun 13;11(6):909. doi: 10.3390/biology11060909. PMID 35741430
- [Background] Reina M, Garcia-Rubio J, Ibanez SJ. Training and Competition Load in Female Basketball: A Systematic Review. Int J Environ Res Public Health. 2020 Apr 12;17(8):2639. doi: 10.3390/ijerph17082639. PMID 32290569
- [Background] Power CJ, Fox JL, Dalbo VJ, Scanlan AT. External and Internal Load Variables Encountered During Training and Games in Female Basketball Players According to Playing Level and Playing Position: A Systematic Review. Sports Med Open. 2022 Aug 19;8(1):107. doi: 10.1186/s40798-022-00498-9. PMID 35984581
- [Background] O Brien J, Browne D, Earls D. The Effects of Different Types of Eccentric Overload Training on Strength, Speed, Power and Change of Direction in Female Basketball Players. J Funct Morphol Kinesiol. 2020 Jul 16;5(3):50. doi: 10.3390/jfmk5030050. PMID 33467266
- [Background] Bouteraa I, Negra Y, Shephard RJ, Chelly MS. Effects of Combined Balance and Plyometric Training on Athletic Performance in Female Basketball Players. J Strength Cond Res. 2020 Jul;34(7):1967-1973. doi: 10.1519/JSC.0000000000002546. PMID 29489714
- [Background] Bright TE, Handford MJ, Mundy P, Lake J, Theis N, Hughes JD. Building for the Future: A Systematic Review of the Effects of Eccentric Resistance Training on Measures of Physical Performance in Youth Athletes. Sports Med. 2023 Jun;53(6):1219-1254. doi: 10.1007/s40279-023-01843-y. Epub 2023 Apr 25. PMID 37097414